CLINICAL TRIAL: NCT04180280
Title: Comparative Effectiveness Trial for Retention, Adherence and Health
Brief Title: Comparative Effectiveness of Brief HIV Care Counseling
Acronym: SWIMS2
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Connecticut (Other)
Collaborators: Mercer University (Other)
Responsible Party: Principal Investigator, Seth Kalichman, Professor, University of Connecticut
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: H14-184GDPH
Record Dates: First submitted 2019-11-25; First posted 2019-11-27 (Actual); Last update posted 2020-05-19 (Actual); Status verified 2020-05

CONDITIONS: HIV/AIDS
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome

STUDY DESIGN:
Intervention Model Description: Behavioral Counseling to Improve HIV Care
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Phone Delivered (Active Comparator): Participants receive 5 sessions of phone-delivered behavioral counseling to improve HIV care.
  Interventions: Behavioral: Behavioral self-regulation Phone counseling to improve HIV care
- Office Delivered (Active Comparator): Participants receive 5 sessions of office-delivered behavioral counseling to improve HIV care.
  Interventions: Behavioral: Behavioral self-regulation Office counseling to improve HIV care

INTERVENTIONS:
Behavioral: Behavioral self-regulation Phone counseling to improve HIV care — Participants receive 5 sessions of behavioral counseling to improve HIV care. Counseling is delivered using phone calls by a trained adherence and care engagement counselor.
  Arms: Phone Delivered
Behavioral: Behavioral self-regulation Office counseling to improve HIV care — Participants receive 5 sessions of behavioral counseling to improve HIV care. Counseling is delivered in clinical care offices s by a trained adherence and care
  Arms: Office Delivered

SUMMARY:
Retention in care and persistent adherence to antiretroviral therapy is necessary for the successful treatment of HIV infection. Alcohol use is known to impede the health care and health outcomes of people living with HIV. The proposed comparative effectiveness study will evaluate the outcomes as well as the facilitators and barriers to implementing a theory-based alcohol counseling intervention that objectively monitors HIV treatment adherence with corrective feedback and increases care engagement delivered by cell phone in resource limited clinical settings.

DETAILED DESCRIPTION:
This application proposes to evaluate the implementation of a theory-based HIV care enhancement and alcohol treatment intervention delivered by cell phone to patients in urban and rural areas. Engagement, retention, and adherence to care are necessary to achieve HIV suppression and antiretroviral therapy (ART) non-adherence can lead to treatment resistant genetic variants of HIV. People living with HIV often experience difficulty sustaining high-levels of treatment adherence and alcohol use is known to impede HIV care. Most factors that interfere with adherence to care are unanticipated and occur between clinical visits, including depression, ART side effects, and substance use. We will conduct a comparative effectiveness study to evaluate the implementation of a cell phone-delivered theory-based alcohol treatment and HIV care adherence counseling intervention. The intervention is grounded in the Behavioral Self-Regulation Model and utilizes brief cell phone counseling that includes monitoring adherence, provider support, and guided corrective feedback as well as interactive text message check-ins. This proactive approach with patients who drink is intended to increase engagement in care and facilitate reductions in drinking thereby improving retention to care and health outcomes. Brief counseling conducted via cell phones allows providers to detect and correct patient slippage from their care plan within a timeframe that can head-off missed appointments, ART non-adherence, and viral resistance. The intervention also includes interactive text (SMS) messaging that begins weekly and tappers off to further enhance engagement in care. Participants are 200 men and 200 women living in high-HIV prevalence remote communities who actively use alcohol and are receiving HIV treatment. Following screening, informed consent, and baseline assessments, participants will be allocated to either (a) the mobile alcohol behavioral self-regulation counseling enhancement to their usual care or (b) routine services provided in their usual care. Participants will be followed for 12-months post-intervention. The primary endpoints are retention to care, medication adherence assessed by unannounced pill counts and HIV RNA (viral load). The study will also evaluate the implementation processes including facilitators and barriers to engagement in care and a cost accounting of resources expended to achieve optimal outcomes. A team of internationally recognized experts in HIV treatment and behavioral research will form a working group to guide an in-depth implementation and cost evaluation. This study will inform the implementation of low-cost evidence-based care retention and adherence interventions in resource limited settings.

ELIGIBILITY:
Inclusion Criteria:

* HIV positive Receiving clinical care New to care Or Returning to care or Not fully engaged in care

Exclusion Criteria:

* HIV Negative Not receiving HIV care

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 400 (Actual)
Dates: Start 2017-06-23 (Actual); Primary Completion 2019-11-01 (Actual); Study Completion 2019-11-01 (Actual)

PRIMARY OUTCOMES:
Engagement in care | 12-months
  Number of participants with clinical appointments attended.

SECONDARY OUTCOMES:
Medication adherence | 12-months
  Percent of medication taken as determined through phone-based medication adherence assessments.

CONTACTS AND LOCATIONS:
Locations (1):
- Share Project, Atlanta, Georgia, United States

IPD SHARING:
Plan to Share IPD: Undecided